CLINICAL TRIAL: NCT04556175
Title: Great Beginnings for Healthy Native Smiles: An Early Childhood Caries Prevention Project
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety concerns for study participants and non-feasibility of enrollment due to the COVID-19 pandemic.
Sponsor: Northern Arizona University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Julie Baldwin, Regents' Professor; Director, Center for Health Equity Research, Northern Arizona University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1396150; 1U01DE028508-01 (NIH)
Record Dates: First submitted 2020-09-01; First posted 2020-09-21 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Early Childhood Caries; Dental Caries
Keywords: child; infant; mothers; pregnant women; dental caries; American Indian, North; motivational interviewing
MeSH Terms: conditions — Dental Caries | interventions — Oral Health

STUDY DESIGN:
Intervention Model Description: Centralized, computer-based group assignment using permuted blocks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Health (Experimental): Motivational interviewing sessions will involve in-person visits by Community Health Workers focused on the mitigation of behavioral risk factors for early childhood caries, with two sessions provided before childbirth and four more sessions at 6, 12, 18 and 24 months after childbirth. Children receive up to 4 fluoride varnish applications during the study. Early cohort of enrollees will be followed up in a 7th visit solely for oral health assessment.
  Interventions: Behavioral: Oral Health
- Healthy Lifestyle (Active Comparator): Didactic educational sessions delivered in-person by Community Health Workers cover nutrition and diet, physical activity, breastfeeding/formula feeding, substance use, mental/emotional health, personal and family goals, prenatal/postpartum health care access, labor and delivery, family support, infant/child care, oral health, and development milestones. Children receive up to 2 fluoride varnish applications during the study. Early cohort enrollees will be followed up in a 7th visit solely for oral health assessment.
  Interventions: Behavioral: Healthy Lifestyle

INTERVENTIONS:
Behavioral: Oral Health — Motivational interviewing for mothers pre-and postpartum; fluoride varnish for infants/children.
  Arms: Oral Health
Behavioral: Healthy Lifestyle — Didactic maternal and child health educational sessions for mothers pre-and postpartum; fluoride varnish for infants/children.
  Arms: Healthy Lifestyle

SUMMARY:
The purpose of this study is to determine whether a bundled best practices oral health intervention utilizing motivational interviewing versus a didactic maternal and child healthy lifestyle intervention will reduce childrens' decayed, missing and/or filled primary tooth surfaces (dmfs) measured over a 2-3 year period.

DETAILED DESCRIPTION:
Early Childhood Caries (ECC) is the most common chronic disease among children. American Indian (AI) children are 4 times more likely to have untreated dental decay than white children. This is a four year parallel group randomized clinical trial evaluating the impact of a bundled best practices oral health intervention on early childhood caries in American Indian children as indicated by the number of decayed, missing and/or filled primary tooth surfaces (dmfs). The intervention is delivered during pregnancy and through child age 24-36 months. The bundled best practices include motivational interviewing with mothers and fluoride varnish applied to the child's teeth. The oral health intervention also includes Tribe-specific individual, social and health needs identified in an earlier formative assessment. The oral health intervention group (n=175 mother-child dyads) will be compared to a group (n=175 mother-child dyads) receiving a standard prenatal/postnatal healthy lifestyle intervention. This comparison Healthy Lifestyle intervention is designed to improve maternal/child health knowledge and also includes Tribe-specific individual, social and health needs identified in an earlier formative assessment. Children in both groups receive some fluoride varnish. All study treatments will be delivered by Community Health Representatives from two Tribal communities in the Western U.S. Children and caregivers will be followed until up to 3 years of age. The primary outcome measure is the average number of decayed, missing and/or filled primary tooth surfaces (dmfs) at the last follow up (24 months for the late enrollment cohort; 30-36 months of age for the early enrollment cohort). Secondary outcomes include 1) the average number of decayed, missing and/or filled primary teeth (dmft) at the last follow up; survey based measures of 2) oral health knowledge; 3) oral health behavior; 4) attitudes towards oral health care; and 5) knowledge of maternal health and child development (e.g., pregnancy related nutrition; breastfeeding; prenatal health).

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Be willing and able to follow study procedures and instructions and be available for the duration of the study
* Be at least 18 years of age (mother)
* Be American Indian or giving birth to an AI child, and living on or near (approximately 100 miles) the Hopi or Crow nations. American Indian status is self-identified-no tribal enrollment verification will be required.
* Be currently pregnant-preferably in month 4 of pregnancy at enrollment but mothers are eligible when 3-7 months pregnant.
* Be willing to participate until the child is age 3
* Mothers of twins will be included, but only one child will be enrolled as the study child.

Exclusion Criteria:

* • Anything that would place the individual at increased risk or preclude the individual's full compliance with, or completion of, the study.

  * Enrolled in other community health interventions that incorporate oral health intervention.
  * A member of the Northern Cheyenne Tribe
  * Living on the Navajo Nation and a member of the Navajo Tribe

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Baldwin, PhD, Principal Investigator — Northern Arizona University
Locations (2):
- United States (2):
  - The Hopi Tribe, Department of Health and Human Services, Kykotsmovi, Arizona
  - Little Big Horn College, Crow Agency, Montana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Health | Healthy Lifestyle
Started | 8 | 8
Completed | 0 | 0
Not Completed | 8 | 8
Not completed — Study terminated due to COVID-19 | 8 | 8

BASELINE CHARACTERISTICS:
Population: Trial was terminated before the outcome measure data were collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Health | Healthy Lifestyle | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There was missing age for one participant
  years
    number analyzed (Participants) | 7 | 8 | 15
    (all) | 28.1 (6.6) | 27.3 (4.6) | 27.7 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 8 | 16
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Decayed, Missing and/or Filled Primary Tooth Surfaces (Dmfs)
Description: For dmfs, there are five surfaces counted on the posterior teeth: facial, lingual, mesial, distal, and occlusal. There are four surfaces counted on anterior teeth: facial, lingual, mesial, and distal. The total tooth count is 20 (8 posterior and 12 anterior) equaling a total of 88 surfaces possible. Each tooth surface will be scored using one of the following mutually exclusive categories; cavitated decayed lesion; filled surface (amalgam); filled surface (non-amalgam); sealed surface; unerupted surface; unable to score. The primary outcome measure is the count of all surfaces scored as cavitated decayed lesion/filled surface/missing due to caries for each individual.
Time Frame: The outcome will be assessed through study completion, child ages 30-36 months for early cohort; 24 months for late cohort. Differential follow up is planned but only the last assessment time point is the primary outcome measure.
Population: Trial was terminated before the outcome measure data were collected
Arm/Group | Oral Health | Healthy Lifestyle
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Decayed, Missing or Filled Primary Teeth (Dmft)
Description: This is a count of the number of teeth with one or more decayed, missing or filled surfaces. This is calculated by counting teeth, rather than tooth surfaces, using the primary outcome assessment (dmfs). If no teeth have been filled or are missing due to disease this outcome is called dt rather than dmft.
Time Frame: The outcome will be assessed through study completion, child ages 30-36 months for early cohort; 24 months for late cohort. Differential follow up is planned but only the last assessment time point is the secondary outcome measure.
Population: Trial was terminated before the outcome measure data were collected
Arm/Group | Oral Health | Healthy Lifestyle
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Oral Health Knowledge of Mothers/Caregivers
Description: Percentage of correct responses to 18 knowledge questions based upon the Basic Research Factors Questionnaire. There are six true/false questions, 8 Likert-type judgements of whether certain behaviors are good for a child's teeth, and 4 multiple choice questions regarding infant/child oral health care.
Time Frame: Oral health knowledge among mothers/caregivers is assessed at Visits 1 (4-7 months pregnant), 4 (child age 12 months) and 6 (child age 24 months).
Population: Trial was terminated before the outcome measure data were collected
Arm/Group | Oral Health | Healthy Lifestyle
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Oral Health Behavior of Mothers/Caregivers
Description: Percentage of correct responses to 12 questions regarding oral health behavior. Eleven are based upon the Basic Research Factors Questionnaire (Wilson et al. Pediatr Dent 2016;38:47-54) and one is based on study-specific question formative assessments. Items include three questions regarding dental health care utilization, seven questions regarding parental involvement in oral health care for self and child and two questions regarding consumption of sweets/sugar.
Time Frame: Oral health behavior among mothers/caregivers is assessed at Visits 4 (child age 12 months) and 6 (child age 24 months).
Population: Trial was terminated before the outcome measure data were collected
Arm/Group | Oral Health | Healthy Lifestyle
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Attitudes Towards Oral Health Care of Mothers/Caregivers
Description: Sum of Likert-type ratings for 14 items. Scores range from 14 (lowest) to 70 (highest) with higher scores representing more favorable attitudes towards child oral health care.
Time Frame: Attitudes towards oral health among mothers/caregivers is assessed at Visits 1 (4-7 months pregnant), 4 (child age 12 months) and 6 (child age 24 months).
Population: Trial was terminated before the outcome measure data were collected
Arm/Group | Oral Health | Healthy Lifestyle
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events were reported by community health worker staff.
Arm/Group | Oral Health | Healthy Lifestyle
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Health (N=8) | Healthy Lifestyle (N=8)
hospitalization (Infections and infestations) | 1 (1) | 0 (0) — Hospitalized for COVID-19
miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — Participant had a miscarriage

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT04556175/Prot_SAP_000.pdf